CLINICAL TRIAL: NCT00625625
Title: Ultrastaging of Early Cancer of the Large Bowel Using Intraoperative Lymphatic Mapping, Sentinel Node Analysis and Blood Testing
Brief Title: Lymphatic Mapping, Sentinel Lymph Node Analysis, and Blood Tests in Detecting and Predicting Early Micrometastases in Patients With Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000586464; JWCI-GULS-CRCSLN-0104
Record Dates: First submitted 2008-02-27; First posted 2008-02-28 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2008-02

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — iso-sulfan blue; Polymerase Chain Reaction; Immunohistochemistry

INTERVENTIONS:
Drug: isosulfan blue
Genetic: polymerase chain reaction
Other: diagnostic laboratory biomarker analysis
Other: immunohistochemistry staining method
Procedure: diagnostic lymphadenectomy
Procedure: therapeutic conventional surgery
Procedure: therapeutic lymphadenectomy

SUMMARY:
RATIONALE: Diagnostic procedures, such as lymph node mapping during surgery and sentinel lymph node biopsy, may help doctors find micrometastases and predict cancer recurrence.

PURPOSE: This phase II trial is studying how well lymph node mapping during surgery together with sentinel lymph node analysis and blood testing work in detecting and predicting early micrometastases in patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the accuracy and sensitivity of intraoperative lymph node mapping with isosulfan blue and sentinal node biopsy (SLN) in patients with colorectal cancer (CRC).
* To compare molecular and immunohistochemical methods for detection of micrometastases in the SLN and primary tumor and evaluate the clinical outcome.
* To evaluate the clinicopathological utility of hematogenous micrometastases in predicting disease recurrence in CRC.

OUTLINE: Patients receive isosulfan blue subserosally around the primary tumor for sentinel lymph node (SLN) identification and SLN(s) are marked. Patients undergo a standard colon resection as planned to include the SLN(s) and regional lymph nodes.

Lymph nodes removed during surgery are analyzed within 30 days after surgery. Routine pathologic analysis (H&E) are performed on all lymph nodes (SLN and non-SLN) removed. Immunohistochemical (IHC) staining for cytokeratin antibodies AE-1/AE-3 or MAK-6 are performed on all lymph nodes negative by H&E. Multimarker PCR (MM PCR) are performed on all SLNs. Blood samples are collected at baseline and then periodically for 4 years for MM PCR to detect circulating tumor cells and standard tumor markers (e.g., CEA).

After surgery, patients are followed every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer as detected by proctosigmoidoscopy, flexible endoscopy, or gastrografin/barium enema
* No evidence of distant metastases by CT scan of the abdomen and pelvis AND chest x-ray or CT scan of the chest performed within 6 weeks prior to enrollment

  * Preoperative CT scans and testing showing non-specific or non-diagnostic (equivocal) abnormalities may be eligible pending intraoperative exploration
* No discovery of distant metastases intra-operatively

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) or Zubrod PS equal to 2
* Life expectancy > 5 years not including the disease/diagnosis of colorectal cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No requirement for emergent surgery (within 2 hours of presentation) to prevent a life-threatening situation or death including:

  * Perforated colon
  * Metabolically significant complete bowel obstruction
  * Massive GI bleeding
  * Occult bleeding or early or partial bowel obstruction not requiring emergent surgery allowed
* No history of Crohn disease, chronic ulcerative colitis, or familial polyposis
* No other malignancy within the past 3 years except for completely resected cervical cancer, skin cancer, or in situ cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* See Patient Characteristics
* No concurrent participation in another research protocol

  * Participation during follow up allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and accuracy of lymphatic mapping in colorectal cancer
Overall survival
Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Shamim Baker — Saint John's Cancer Institute